CLINICAL TRIAL: NCT03689712
Title: ROMAN: Reduction in Oral Mucositis With Avasopasem Manganese (GC4419) - Phase 3 Trial in Patients Receiving Chemoradiotherapy for Locally-Advanced, Non-Metastatic Head and Neck Cancer
Brief Title: ROMAN: Phase 3 Trial Investigating the Effects of GC4419 on Radiation Induced Oral Mucositis in Head/Neck Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GTI-4419-301
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Results first posted 2023-04-13 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Oral Mucositis
Keywords: Oral Mucositis; Superoxide Dismutase Mimetic; Cisplatin; Intensity-Modulated Radiation Therapy; Chemoradiation; OM; IMRT; Head and Neck Cancer; Squamous Cell Carcinoma; SCC; Oral Cavity; Oropharnyx; Mouth Sores; avasopasem mangenese
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms; Carcinoma, Squamous Cell; Oral Ulcer | interventions — avasopasem manganese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GC4419 (avasopasem manganese) 90 mg (Experimental)
  Interventions: Drug: GC4419 90mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GC4419 90mg — 60 minute IV infusion
  Other Names: avasopasem manganese
  Arms: GC4419 (avasopasem manganese) 90 mg
Drug: Placebo — 60 minute IV infusion
  Arms: Placebo

SUMMARY:
The purpose of the phase 3, clinical study is to determine if GC4419 (avasopasem manganese) administered prior to intensity-modulated radiation therapy (IMRT) reduces the severity of radiation induced oral mucositis in patients who have been diagnosed with locally advanced, non-metastatic squamous cell carcinoma of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

* squamous cell carcinoma of the head and neck
* treatment plan to receive IMRT delivered as single daily fractions of 2.0 to 2.2 Gy with a cumulative radiation dose of 60-72 Gy
* Treatment plan to receive standard cisplatin monotherapy
* Age 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate hematologic, renal and liver function
* Negative serum pregnancy test
* Use of effective contraception

Exclusion Criteria:

* Tumor of the lips, larynx, hypopharynx, nasopharynx, sinuses, or salivary glands
* Metastatic disease
* Prior radiotherapy to the region of the study cancer or adjacent anatomical
* Prior induction chemotherapy
* Receiving any approved or investigational anti-cancer agent other than those provided for in this study
* Concurrent participation in another interventional clinical study
* Inability to eat soft solid food at baseline
* Malignant tumors other than HNC within the last 5 years
* Active infectious disease excluding oral candidiasis
* Presence of oral mucositis at baseline
* Known history of HIV or active hepatitis B/C
* Female patients who are pregnant or breastfeeding
* Known allergies or intolerance to cisplatin and similar platinum-containing compounds
* Requirement for concurrent treatment with nitrates or other drugs that may create a risk for a precipitous decrease in blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2023-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gene Kennedy, MD, Study Chair — Galera Therapeutics
Locations (97):
- United States (86):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Fowler Family Center for Cancer, Jonesboro, Arkansas
  - The Oncology Institute of Hope & Innovation, Corona, California
  - Chan Soon-Shiong Institute for Medicine, Costa Mesa, California
  - Long Beach Veteran Affairs Healthcare System, Long Beach, California
  - USC Norris Cancer Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Clinical Trials and Research Associates, Inc., Montebello, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Compassionate Cancer Care, Riverside, California
  - Sharp Clinical Oncology Research, San Diego, California
  - The Oncology Institute of Hope & Innovation, Whittier, California
  - Dignity Health Research Institute, Woodland, California
  - St. Mary's Hospital Regional Medical Center, Grand Junction, Colorado
  - Bay Pines VA HealthCare System, Bay Pines, Florida
  - Boca Raton Regional Hospital, Lynn Cancer Institute, Boca Raton, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - BRCR Global, Plantation, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - IACT Health, Columbus, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - SwedishAmerican Regional Cancer Center, Rockford, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - The University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Appalachian Regional Healthcare, INC., Hazard, Kentucky
  - University of Louisville/James Graham Brown Cancer Center, Louisville, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - MetroWest Medical Center, Framingham, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Minneapolis VA Healthcare System, Minneapolis, Minnesota
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - Henry Ford Allegiance Health Hematology Oncology, Jackson, Mississippi
  - Ellis Fischel Cancer Center - University of Missouri, Columbia, Missouri
  - Delbert Day Cancer Institute, Phelps County Regional Medical Center, Rolla, Missouri
  - Mosaic Life Care/Heartland Regional Medical Center, Saint Joseph, Missouri
  - Cox Medical Center, Springfield, Missouri
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Benefis Sletten Cancer institute, Great Falls, Montana
  - CHI Health St. Francis, Grand Island, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Exeter Hospital, Exeter, New Hampshire
  - Hunterdon Hematology Oncology, LLC, Flemington, New Jersey
  - Summit Medical Group, Florham Park, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - New York Oncology Hematology, P.C., Albany, New York
  - NY Cancer and Blood Specialists, East Setauket, New York
  - New York- Presbyterian Queens/ Weill Cornell, Flushing, New York
  - Wilmot Cancer Institute - Univeristy of Rochester, Rochester, New York
  - School of Dental Medicine at East Carolina University, Greenville, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Summa Health, Akron, Ohio
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Willamette Valley Cancer Institue and Research Center, Eugene, Oregon
  - VA Portland Health Care System, Portland, Oregon
  - St. Luke's Hospital Cancer Center, Easton, Pennsylvania
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Anmed Health Cancer Center, Anderson, South Carolina
  - Charleston Cancer Center, Charleston, South Carolina
  - St. Francis Cancer Center, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Mountain States Health Alliance Research Dept, Johnson City, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Texas Oncology - Beaumont Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology- Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Denton South, Denton, Texas
  - Texas Oncology - El Paso Cancer Treatment Center, El Paso, Texas
  - SAMMC, Fort Sam Houston, Texas
  - Texas Oncology-McAllen, McAllen, Texas
  - Texas Oncology - McKinney, McKinney, Texas
  - Texas Oncology, Plano West, Plano, Texas
  - Baylor Scott & White- Round Rock, Round Rock, Texas
  - Texas Oncology - Sugar Land, Sugar Land, Texas
  - Texas Oncology - Waco, Waco, Texas
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Roanoke, Virginia
  - Providence Regional Cancer Partnership, Everett, Washington
  - Cancer Care Northwest, Spokane, Washington
  - West Virginia University, Morgantown, West Virginia
- Canada (10):
  - BC Cancer Center - Vancouver, Vancouver, British Columbia
  - CIUSS de L'Est-de-I'lle de Montreal - Hopital Maisonneuve- Rosemont, Montreal, Quebec
  - McGill University Health Center- Cedars Cancer Center, Montreal, Quebec
  - CHU de Quebec - Universite Laval, Québec, Quebec
  - Centre Intégré Universitaire de Santé et de Services Sociaux du Saguenay-Lac-Saint-Jean, Chicoutimi
  - Northeast Cancer Centre of Health Sciences North, Greater Sudbury
  - Juravinski Cancer Centre, Hamilton
  - Centre Hospitalier Universitaire de Montreal (CHUM), Montreal
  - Jewish General Hospital, Montreal
  - Centre Intégré Universitaire de Santé et de Services Sociaux de la Mauricie et du Centre du Québec, Trois-Rivières
- Clinical Research Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson CM, Lee CM, Kelley JR, et al. ROMAN: Phase 3 trial of avasopasem manganese (GC4419) for severe oral mucositis (SOM) in patients receiving chemoradiotherapy (CRT) for locally advanced, nonmetastatic head and neck cancer (LAHNC). Journal of Clinical Oncology 2022 40:16_suppl, 6005-6005
- [Background] Saunders D, Lee C, Kelley J, et al. ROMAN: Phase 3 trial of avasopasem to reduce chemoradiotherapy (CRT)-related severe oral mucositis (SOM) in patients with head and neck cancer (HNC). Support Care Cancer 30 (Suppl 1), 1-207 (2022).
- [Derived] Anderson C, Lee CM, Kelley JR, Walker GV, Dunlap NE, Bar-Ad VC, Miller DA, King VJ, Peddada AV, Ciuba DF, Vincent F, Muzyka BC, Gillespie-Twardy AL, Sonis ST, Holmlund J, Beardsley RA, Kennedy EP, Saunders D. Avasopasem manganese treatment for severe oral mucositis from chemoradiotherapy for locally advanced head and neck cancer: phase 3 randomized controlled trial (ROMAN). EClinicalMedicine. 2025 Oct 8;89:103539. doi: 10.1016/j.eclinm.2025.103539. eCollection 2025 Nov. PMID 41127563
- [Derived] Squillace S, Salvemini D. Nitroxidative stress in pain and opioid-induced adverse effects: therapeutic opportunities. Pain. 2022 Feb 1;163(2):205-213. doi: 10.1097/j.pain.0000000000002347. No abstract available. PMID 34145168
- [Derived] Anderson CM, Lee CM, Saunders DP, Curtis A, Dunlap N, Nangia C, Lee AS, Gordon SM, Kovoor P, Arevalo-Araujo R, Bar-Ad V, Peddada A, Colvett K, Miller D, Jain AK, Wheeler J, Blakaj D, Bonomi M, Agarwala SS, Garg M, Worden F, Holmlund J, Brill JM, Downs M, Sonis ST, Katz S, Buatti JM. Phase IIb, Randomized, Double-Blind Trial of GC4419 Versus Placebo to Reduce Severe Oral Mucositis Due to Concurrent Radiotherapy and Cisplatin For Head and Neck Cancer. J Clin Oncol. 2019 Dec 1;37(34):3256-3265. doi: 10.1200/JCO.19.01507. Epub 2019 Oct 16. PMID 31618127

RESULTS

PARTICIPANT FLOW:
Groups:
- GC4419 (Avasopasem Manganese) 90 mg: GC4419 (avasopasem manganese): 60 minute IV infusion
Period: Overall Study
Arm/Group | GC4419 (Avasopasem Manganese) 90 mg | Placebo
Started | 270 | 185
Intent to Treat Population (Intent-to-Treat (ITT) population includes all randomized subjects who received at least one dose of GC4419/Placebo, with the exception of the 28 subjects whose treatment course was discontinued during the Sponsor's voluntary suspension of dosing.) | 241 | 166
Completed | 105 | 74
Not Completed | 165 | 111
Not completed — Adverse Event | 1 | 0
Not completed — Death | 20 | 10
Not completed — Lost to Follow-up | 6 | 6
Not completed — Other | 1 | 0
Not completed — Patient Non-Compliance | 0 | 1
Not completed — Withdrawal by Subject | 20 | 4
Not completed — Patients Continuing in Long Term Follow Up | 88 | 71
Not completed — Randomized but not Treated | 13 | 7
Not completed — Subject Dosing Suspended due to Product Issue | 16 | 12

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population includes all randomized subjects who received at least one dose of GC4419/Placebo, with the exception of the 28 subjects whose treatment course was discontinued during the Sponsor's voluntary suspension of dosing.
Groups:
- GC4419 (Avasopasem Manganese): GC4419 (avasopasem manganese): 60 minute IV infusion
- Total: Total of all reporting groups
Arm/Group | GC4419 (Avasopasem Manganese) | Placebo | Total
Number analyzed (Participants) | 241 | 166 | 407
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 163 | 111 | 274
  >=65 years | 78 | 55 | 133
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 17 | 56
  Male | 202 | 149 | 351
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 1 | 9
  Not Hispanic or Latino | 222 | 160 | 382
  Unknown or Not Reported | 11 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 10 | 2 | 12
  White | 219 | 158 | 377
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  Canada | 33 | 24 | 57
  United States | 208 | 142 | 350

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Severe Oral Mucositis
Description: Cumulative incidence of severe oral mucositis is defined as the proportion of subjects with any occurrence of WHO Grade 3 to 4 OM, during the Study Treatment Period. Incidence of severe OM is defined as any occurrence of WHO Grade 3 or 4 OM through the last IMRT fraction after the start of IMRT. Incidence was imputed using multiple imputation for subjects with incomplete follow-up for severe OM through 60 Gy who did not have an occurrence of severe OM before the last IMRT fraction.
Time Frame: From the first IMRT fraction through the end of the study treatment period (completion of study drug administration, IMRT and chemotherapy), which is estimated to be 7 weeks.
Population: The Intent to treat population consisted of all randomized subjects who received at least 1 dose of avasopasem manganese or placebo (with the exception of subjects whose treatment course was discontinued due to the sponsor's voluntary suspension of dosing)
Measure: Number; unit: percentage of patients
Groups:
- GC4419 (Avasopasem Manganese) 90mg: GC4419: 60 minute IV infusion
Arm/Group | GC4419 (Avasopasem Manganese) 90mg | Placebo
Number analyzed (Participants) | 241 | 166
percentage of patients | 53.8 | 64.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first dose of GC4419 (avasopasem manganese)/Placebo until 30 days following the last dose of GC4419 (avasopasem manganese)/Placebo, IMRT, or chemotherapy (whichever was later). Timeframe for collection of adverse events was approximately 10 weeks
Arm/Group | GC4419 (Avasopasem Manganese) 90 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 20/241 | 10/166
Serious Adverse Events (participants affected / at risk) | 81/241 | 52/166
Other Adverse Events (participants affected / at risk) | 240/241 | 166/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GC4419 (Avasopasem Manganese) 90 mg (N=241) | Placebo (N=166)
Febrile Neutropenia (Blood and lymphatic system disorders) | 15 (17) | 8 (9)
Dehydration (Metabolism and nutrition disorders) | 7 (8) | 3 (3)
Sepsis (Infections and infestations) | 4 (4) | 4 (5)
Failure to Thrive (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 5 (7)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Pyrexia (General disorders) | 6 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 6 (6)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 2 (4)
Lung Infection (Infections and infestations) | 2 (2) | 2 (2)
Asethenia (General disorders) | 1 (1) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Device Malfunction (Product Issues) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hepatitis viral (Infections and infestations) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Weight Decreased (Investigations) | 0 (0) | 2 (2)
Abdominal Wall Abscess (Infections and infestations) | 1 (1) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Bactaraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Corona Virus Infection (Infections and infestations) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Device Occulsion (Product Issues) | 1 (1) | 0 (0)
Device Related Infection (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Euglycaemic Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gastrostomy Tube Removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastrostomy Tube Site Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lipase Increased (Investigations) | 1 (1) | 0 (0)
Metastases to Peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Neutropenic Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Staphylococcal Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Stoma Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GC4419 (Avasopasem Manganese) 90 mg (N=241) | Placebo (N=166)
Lymphopenia (Blood and lymphatic system disorders) | 212 (465) | 155 (329)
Nausea (Gastrointestinal disorders) | 207 (449) | 137 (319)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 146 (280) | 113 (251)
Fatigue (General disorders) | 170 (278) | 124 (238)
Constipation (Gastrointestinal disorders) | 154 (236) | 102 (194)
Radiation Skin Injury (Injury, poisoning and procedural complications) | 126 (222) | 104 (181)
Vomiting (Gastrointestinal disorders) | 135 (259) | 77 (137)
Weight Decreased (Investigations) | 116 (222) | 80 (148)
Paresthesia (Nervous system disorders) | 36 (212) | 15 (41)
Dysgeusia (Nervous system disorders) | 137 (192) | 119 (167)
Dry Mouth (Gastrointestinal disorders) | 129 (163) | 104 (152)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the proposed manuscript (or other document) for publication, presentation or other disclosure must be forwarded to the sponsor not less than 30 days prior to submission or presentation and the Principal Investigator shall comply with Sponsor's requests to delete or revise references to Confidential Information and consider all other comments of Sponsor in good faith.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT03689712/Prot_SAP_000.pdf